CLINICAL TRIAL: NCT03882619
Title: Effectiveness of Using Calligraphic Activity to People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Jianan Psychiatric Center, Ministry of Health and Welfare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 19-001
Record Dates: First submitted 2019-03-13; First posted 2019-03-20 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calligraphy group (Experimental)
  Interventions: Behavioral: Calligraphy
- Treatment-as-usual group (No Intervention)

INTERVENTIONS:
Behavioral: Calligraphy — Participants will (1) detect the emotion him or herself; (2) do the calligraphy activity by writing positive terms (e.g., peace, life); (3) detect emotion again; (4) share the experience with group members.
  Arms: Calligraphy group

SUMMARY:
To examine the effects of calligraphy activity on symptoms, attention, emotion, and quality of life in people with schizophrenia. We hypothesized that through a six-month intervention using calligraphy activity, people with schizophrenia will have their symptoms decreased, attention improved, emotion enhanced, and quality of life increased. This study will adopt single-blind, randomized controlled trial, and 160 people with schizophrenia will be recruited in this study. They will be randomly assigned to either a calligraphy activity group (treatment group; n=80) or an occupational activity group (control group; n=80). Participants will complete assessments at pretest, posttest, and 3-month follow-up using the following instruments: Positive and Negative Syndrome Scale (PANSS), Chu's Attention Test, The Taiwanese version of Montreal Cognitive Assessment (MoCA-T), WHO questionnaire on the Quality of Life, Brief Form (WHOQOL-BREF), and Chinese Depression Anxiety Stress Scales(DASS21).

ELIGIBILITY:
Inclusion Criteria:

* Inpatients
* With diagnosis of schizophrenia or schizoaffective disorder
* Not in acute stage
* Voluntarily participate

Exclusion Criteria:

* Severe cognition level or intellectual disability that prevent from participation
* Severe behavioral problems and symptoms that prevent from participation
* People with blindness

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in emotion | Changes from baseline, end of study (3 months after baseline), and 6 months after baseline
  Emotion is assessed using self-report of Chinese Depression Anxiety Stress Scale. The scale includes three subscales: depression (score range 0-21; higher score indicates higher depression), anxiety (score range 0-21; higher score indicates higher anxiety), and stress (score range 0-21; higher score indicates higher stress).
Changes in attention | Changes from baseline, end of study (3 months after baseline), and 6 months after baseline
  Attention is assessed using Chu's Attention Test. The test contains 200 items and is assessed in 10 minutes with two scores calculated: correct number (answered number-number of error answer); rate of correct number (correct number divided by answered number). Higher scores in correct number and rate of correct number indicate better attention.
Changes in syndrome | Changes from baseline, end of study (3 months after baseline), and 6 months after baseline
  Symptoms are assessed using Positive and Negative Syndrome Scale. The scale includes three subscales: positive symptom (score range 7-49; higher score indicates more positive symptoms), negative symptoms (score range 7-49; higher score indicates more negative symptoms), and general psychopathology (score range 16-112; higher score indicates more general symptoms).
Changes in cognition | Changes from baseline, end of study (3 months after baseline), and 6 months after baseline
  Cognition is assessed using Taiwanese version of Montreal Cognitive Assessment. The score range of the scale is between 0 and 30, a higher score indicates better cognition.
Changes in quality of life | Changes from baseline, end of study (3 months after baseline), and 6 months after baseline
  Quality of life is assessed using WHO questionnaire on the Quality of Life, Brief Form. The scale includes four subscales: physical (score range 4-20; higher score indicates better physical quality of life); psychological (score range: 4-20; higher score indicates better psychological quality of life); social (score range: 4-20; higher score indicates better social quality of life); environment (score range: 4-20; higher score indicates better environment quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Jianan Psychiatric Center, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang WY, Tsang HWH, Wang SM, Huang YC, Chen YC, Cheng CH, Chen CY, Chen JS, Chang YL, Huang RY, Lin CY, Potenza MN, Pakpour AH. Effectiveness of using calligraphic activity to treat people with schizophrenia: a randomized controlled trial in Southern Taiwan. Ther Adv Chronic Dis. 2022 Mar 11;13:20406223221080646. doi: 10.1177/20406223221080646. eCollection 2022. PMID 35295614